CLINICAL TRIAL: NCT07229976
Title: Clinical Efficacy of Thumbtack Needle for Chronic Insomnia in Perimenopausal and Menopausal Women: A Multicenter Randomized Controlled Trial
Brief Title: Clinical Efficacy of Thumbtack Needle for Chronic Insomnia in Perimenopausal and Menopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dongmei Huang, Dr, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-IRB202510056
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Insomnia During Perimenopause and Menopause

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thumbtack needle group (Experimental): The subject received thumbtack needle
  Interventions: Other: thumbtack needle
- Placebo thumbtack needle group (Other): The subject received placebo thumbtack needle
  Interventions: Other: placebo thumbtack needle

INTERVENTIONS:
Other: thumbtack needle — The treatment acupoints include bilateral Anmian Acupoint, bilateral Taichong acupoints, bilateral Neiguan acupoints, bilateral Sanyinjiao (SP6), and bilateral Zusanli (ST36) and Danzhong acupoints, a total of 11 acupoints. After 3 days of thumbtack needle retention, the patient went to the hospital where the doctor removed the thumbtack needle, disinfected the local skin, and received the next needle treatment. The patient received treatment twice a week (6 days) and rested for 1 day before continuing with the next treatment.
  Arms: thumbtack needle group
Other: placebo thumbtack needle — The placebo thumbtack needle group selected acupoints that were the same as the thumbtack needle group. Bilateral sleeping acupoints, bilateral Taichong acupoints, bilateral Neiguan acupoints, bilateral Sanyinjiao (SP6), bilateral Zusanli (ST36), and Danzhong acupoints are all treated with comforting acupressure.where the doctor removed the placebo thumbtack needle, disinfected the local skin, and received the next placebo thumbtack needle needle. The patient received treatment twice a week (6 days) and rested for 1 day before continuing with the next treatment.
  Arms: Placebo thumbtack needle group

SUMMARY:
A multicenter, randomized, controlled, blinded clinical trial was conducted to evaluate the effects of thumbtack needle on sleep in patients with chronic insomnia during perimenopause and menopause. Randomly divided into a treatment group and a control group using the central area method, with 99 patients in each group. The treatment group received thumbtack needle treatment, while the control group received placebo thumbtack needle treatment. The treatment course for both groups was 4 weeks.

ELIGIBILITY:
Diagnostic criteria for perimenopause and menopause:

* Perimenopausal period: a period of time from one year before the last menstrual period to the first year after the last menstrual period. Having at least one menstrual period in the past 12 months, or being under 55 years old, undergoing hysterectomy or endometrial ablation, but not bilateral oophorectomy;
* Menopause: No menstruation in the past 12 months, or bilateral oophorectomy, or age 55 years or older, who has undergone hysterectomy or endometrial ablation;

Diagnostic criteria for chronic insomnia:

●The diagnostic criteria for insomnia in the third edition of the International Classification of Sleep Disorders (ICSD-3) of the American Academy of Sleep Medicine (all criteria A to F must be met).

Inclusion Criteria:

* Women aged 40 to 65 who meet the diagnostic criteria for perimenopause and menopause mentioned above;
* Evaluate ISI score ≥ 12 points through a scale;
* Meets the diagnostic criteria for chronic insomnia mentioned above, i.e. ICSD-3 meets both criteria A to F;
* Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

Patients who meet any of the following conditions will not be included;

* Use hormone replacement therapy, anti anxiety drugs, antidepressants, or medications to improve insomnia within one month;
* Individuals with a history of diagnosed sleep disorders before menopause;
* Combined with other sleep disorders such as obstructive sleep apnea, restless leg syndrome, etc;
* Patients with malignant tumors, especially estrogen dependent tumors (such as breast cancer and endometrial cancer);
* Recent (within 6 months) history of myocardial infarction, stroke, venous thrombosis, etc;
* Patients with mental illnesses, such as severe depression and uncontrolled schizophrenia;
* Serious disorder of endocrine system, such as uncontrolled hyperthyroidism, diabetes ketoacidosis, etc
* Patients with coagulation disorders, such as hemophilia, long-term use of anticoagulants (warfarin, aspirin, etc.), etc;
* Long term alcohol consumption history (more than 5 years, daily alcohol consumption exceeding 12 taels, not quitting drinking);
* Engaged in night shift work (>3 times a week);
* Individuals with infections, ulcers, burns, rashes, or scars at acupoints;
* Previously received acupuncture treatment;
* I do not agree to sign the informed consent form for this study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 2 weeks, 4 weeks, 2 months
  The Insomnia Severity Index (ISI) is a self-assessment tool used to evaluate the severity of insomnia. The ISI scale consists of 7 items, each rated on a scale of 0-4, with a total score range of 0-28 points. Evaluate the difference in scores between the Insomnia Severity Index (ISI) scale at the end of week 2 and week 4 and baseline ISI scores. Evaluate the difference between the ISI score at the end of the 4-week follow-up period and baseline ISI scores .

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | 4 weeks, 2 months
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used sleep quality assessment tool internationally. Evaluate the difference between the PSQI score at the end of week 4 and the baseline PSQI score. Evaluate the difference between the PSQI score at the end of the 4-week follow-up and the baseline PSQI score.
Epworth Sleepiness Scale | 4 weeks, 2 months
  The Epworth Sleepiness Scale (ESS) is a self-assessment tool used to evaluate an individual's level of daytime sleepiness. Evaluate the difference between the ESS score at the end of week 4 and the baseline ESS score. Evaluate the difference between ESS score at the end of 4 weeks of follow-up and baseline ESS score .
Fatigue Severity Scale | 4 weeks, 2 months
  The Fatigue Severity Scale (FSS) is currently one of the most commonly used scales for assessing fatigue symptoms in clinical practice. Assess the difference between FSS score at the end of week 4 and baseline FSS score . Evaluate the difference between FSS score at the end of 4 weeks of follow-up and baseline FSS score .
Zung Self Rating Anxiety Scale | 4 weeks, 2 months
  The Zung Self Rating Anxiety Scale (SAS) is used to assess the severity of an individual's anxiety symptoms over the past week. Evaluate the difference between the SAS score at the end of week 4 and the baseline SAS score. Evaluate the difference between SAS score at the end of 4 weeks of follow-up and baseline SAS score .
Zung Self Rating Depression Scale | 4 weeks, 2 months
  The Zung Self Rating Depression Scale (SDS) is currently one of the most widely used self-assessment scales for depression. Evaluate the difference between SDS score at the end of week 4 and baseline SDS score. Evaluate the difference between SDS score at the end of 4 weeks of follow-up and baseline SDS score .
Sleep efficiency | 2 weeks，4 weeks and 2 months
  Sleep efficiency refers to the ratio of actual sleep time to bed rest time. Evaluate the difference between sleep efficiency at the end of week 2 and week 4 and baseline sleep efficiency. Evaluate the difference between sleep efficiency at the end of 4 weeks of follow-up and baseline sleep efficiency.
wake-up time after sleep onset | 2 weeks, 4 weeks and 2 months
  Assess the difference between the wake-up time after sleep onset at the end of week 2 and week 4, and the wake-up time after baseline sleep onset. Evaluate the difference between the wake-up time after sleep onset at the end of 4 weeks of follow-up and the wake-up time after baseline sleep onset.
the number of awakenings per night | 2 weeks, 4 weeks and 2 months
  Evaluate the difference between the number of awakenings per night at the end of week 2 and week 4 compared to the baseline number of awakenings per night. Evaluate the difference between the number of awakenings per night at the end of 4 weeks of follow-up and the baseline number of awakenings per night.
The latent period of sleep onset | 2 weeks, 4 weeks and 2 months
  The latent period of sleep onset refers to the time it takes from getting ready to sleep to actually entering a state of sleep. Evaluate the difference between the sleep onset latency at the end of week 2 and week 4 and the baseline sleep onset latency. Evaluate the difference between the sleep onset latency at the end of 4 weeks of follow-up and the baseline sleep onset latency.
Total sleep time | 2 weeks, 4 weeks and 2 months
  Total sleep time refers to the total duration of continuous or intermittent sleep that an individual experiences within a certain period of time (usually 24 hours). Evaluate the difference between the total sleep time at the end of week 2 and week 4 and the baseline total sleep time. Evaluate the difference between the total sleep time at the end of the 4-week follow-up and the baseline total sleep time.
the average wake-up time | 2 weeks, 4weeks and 2 months
  Evaluate the difference between the average wake-up time at the end of week 2 and week 4 and the baseline average wake-up time. Evaluate the difference between the average wake-up time at the end of the 4-week follow-up and the baseline average wake-up time.
Corticotropin-Releasing Hormone | 4 weeks
  Corticotropin Releasing Hormone (CRH) is a peptide hormone secreted by the hypothalamus. Evaluate the difference in serum CRH concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
Norepinephrine | 4 weeks
  Norepinephrine is both a neurotransmitter and a hormone. Evaluate the difference in serum Norepinephrine concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
Adrenaline | 4 weeks
  Adrenaline is a hormone and neurotransmitter secreted by the adrenal medulla. Evaluate the difference in serum Adrenaline concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
5-hydroxytryptamine | 4 weeks
  5-hydroxytryptamine (5-HT), also known as serotonin, is an important monoamine neurotransmitter that plays a crucial role in the physiological and psychological functions of the human body. Evaluate the difference in serum 5-HT concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
Gamma aminobutyric acid | 4 weeks
  Gamma aminobutyric acid (GABA) is a non protein amino acid widely present in the human body, animals, and plants, and is also an important inhibitory neurotransmitter in the central nervous system. Evaluate the difference in serum GABA concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
Dopamine | 4 weeks
  Dopamine is an important neurotransmitter that has a wide range of effects on human physiological and psychological functions. Evaluate the difference in serum Dopamine concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
Melatonin | 4 weeks
  Melatonin is an endogenous hormone secreted by the pineal gland of the human brain. Evaluate the difference in serum melatonin concentration between the thumbtack needle group and the placebo thumbtack needle group at the end of week 4.
β - endorphin | 4 weeks
  Evaluate the difference in serum β - endorphin concentration between the placebo group and the placebo group at the end of week 4.
insomnia remission rate | 4 weeks
  The proportion of patients who no longer meet the diagnosis of insomnia after treatment among those receiving insomnia treatment. The diagnosis of insomnia refers to the International Classification of Sleep Disorders, ICSD-3
Insomnia Treatment Response Rate | 4 weeks
  The proportion of patients receiving insomnia treatment whose Insomnia Severity Index score decreased by 8 or more points after treatment